CLINICAL TRIAL: NCT03251443
Title: Single Center, Single Arm, Open Study, to Explore and Evaluate Treatment of Apatinib in Patients With Advanced Intrahepatic Cholangiocarcinoma
Brief Title: A Study of Second-line Treatment With Apatinib in Patients With Advanced Intrahepatic Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-1392
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2019-07

CONDITIONS: Intrahepatic Cholangiocarcinoma; Second-line Treatment
MeSH Terms: conditions — Cholangiocarcinoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib (Experimental): A molecular targeted anti-tumor drugs. Small molecule vascular endothelial growth factor receptor 2 inhibitor.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — 500mg, once a day, oral of each 28 day cycle. Number of cycle: until progression or unacceptable toxicity develops.
  Other Names: Apatinib mesylate tablets

SUMMARY:
The purpose of this study is to explore the efficacy and safety of second-line treatment of apatinib in advanced intrahepatic cholangiocarcinoma patients and evaluate drug safety, progression free and overall survival. The primary endpoint of this study is objective response rate (ORR), disease control rate (DCR) and progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic or cytologic diagnosis of intrahepatic cholangiocarcinoma with stage IV;
* Have progressed after systematic chemotherapy/target therapy, or cannot tolerated with first-line treatment;
* The previous treatment and the present trial registration must be at least 2 weeks apart, and they must have recovered from any toxicity of a previous treatment;
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1;
* Eastern Cooperative Oncology Group performance score (ECOG): 0-2;
* Life expectancy of at least 12 weeks;
* Subjects who understand and voluntarily signed a written informed consent form.

Exclusion Criteria:

* Previous locoregional therapy within 4 weeks prior to enrollment.
* Diagnosed with hepatocellular carcinoma, mixed cell carcinoma and fibrolamellar hepatocellular carcinoma.
* History of other malignancy within 5 years except for non-melanoma skin cancer, cervix in situ carcinoma.
* Prepared for liver transplantation.
* Patients with contraindications (active bleeding, ulcers, intestinal perforation, intestinal obstruction, within 30 days after major surgery, uncontrolled high blood pressure medication, III-IV level cardiac insufficiency, severe liver and kidney dysfunction).
* A previous history of Interstitial pulmonary disease, drug-induced interstitial disease, radiation pneumonitis requiring hormonal therapy or active interstitial lung disease with any clinical evidence.
* Use of CYP3A4 inhibitor within 7 days or CYP3A4 inducer within 12 days prior to enrollment.
* Patients with central nervous system metastases or brain metastasis
* Previous definite diagnosis of neuropsychiatric disturbances, including epilepsy or dementia.
* Pregnant or lactating women.
* Patients with bone metastasis received palliative radiation within 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | six months
  A duration from the date of initial treatment with apatinib to disease progression (as defined by RECIST) or death.
Objective Response Rate (ORR) | one year
Disease Control Rate (DCR) | one year

SECONDARY OUTCOMES:
Overall Survival (OS) | two years
  Overall survival (OS) was calculated from the date of initial treatment with apatinib to the date of death due to any cause
Incidence of Treatment-Emergent Adverse Event | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hai-tao Zhao, Study Chair — Peking Union Medical College Hospital (PUMCH)
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China